CLINICAL TRIAL: NCT01368237
Title: Dynamic Myocardial Perfusion Imaging by 320 Multidetector Computed Tomography
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 210/R/CAR/11
Record Dates: First submitted 2011-06-06; First posted 2011-06-07 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2014-10

CONDITIONS: Coronary Heart Disease
Keywords: Computed tomography; Myocardial perfusion; Coronary heart disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Patients awaiting invasive coronary angiography
  Interventions: Radiation: Computed tomography scan

INTERVENTIONS:
Radiation: Computed tomography scan — Computed tomography will be performed using a 320 multidetector computed tomography scanner and may include coronary calcium score, coronary angiography and imaging of myocardial perfusion, function and viability.

SUMMARY:
Recent advances in technology have resulted in the development of scanners that can image the heart blood vessels within 10 to 20 minutes but without the need for admission to hospital or insertion of catheters. Further advances in technology allow the visualisation of both the blood vessels and the supply of blood to the heart muscle. Here we propose to assess the latest and most powerful computed tomography scanner and compare it to magnetic resonance and conventional coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

* referred for invasive coronary angiography because of suspected coronary heart disease

Exclusion Criteria:

* inability or unwillingness to undergo computed tomography or magnetic resonance imaging
* renal failure (serum creatinine >200 micromol/L or estimated glomerular filtration rate <30 mL/min)
* hepatic failure
* allergy to iodinated contrast or gadolinium
* pregnancy
* contraindication to adenosine infusion
* inability to give informed consent
* inability to perform fractional flow reserve during invasive coronary angiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients awaiting invasive coronary angiography
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2006-05; Primary Completion 2014-06 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Myocardial perfusion defects defined qualitatively by trained observers and quantitatively by computer software | 1 month
  The primary outcome measure is to establish whether 320-multidetector computed tomography can identify myocardial perfusion defects as compared to the gold standards of 3Tesla magnetic resonance imaging and fractional flow reserve measured during invasive coronary angiography.

SECONDARY OUTCOMES:
Identification of regional wall motion abnormalities qualitatively by trained observers | 1 month
  Our secondary outcome measures are to assess the performance of 320-multidetector computed tomography in the detection of regional wall motion abnormalities in comparison to those obtained with 3Tesla cardiac magnetic resonance imaging.
Identification of infarction qualitatively by trained observers | 1 month
  Our secondary outcome measures are to assess the performance of 320-multidetector computed tomography in the detection of infarction in comparison to those obtained with 3Tesla cardiac magnetic resonance imaging.
Identification of regional wall motion abnormalities quantitatively by computer software | 1 month
  Our secondary outcome measures are to assess the performance of 320-multidetector computed tomography in the detection of regional wall motion abnormalities in comparison to those obtained with 3Tesla cardiac magnetic resonance imaging.
Identification of infarction qualitatively by computer software | 1 month
  Our secondary outcome measures are to assess the performance of 320-multidetector computed tomography in the detection of infarction in comparison to those obtained with 3Tesla cardiac magnetic resonance imaging.

CONTACTS AND LOCATIONS:
Overall Officials: David E Newby, Principal Investigator — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Scotland, United Kingdom

REFERENCES:
- [Derived] Papanastasiou G, Williams MC, Dweck MR, Alam S, Cooper A, Mirsadraee S, Newby DE, Semple SI. Quantitative assessment of myocardial blood flow in coronary artery disease by cardiovascular magnetic resonance: comparison of Fermi and distributed parameter modeling against invasive methods. J Cardiovasc Magn Reson. 2016 Sep 13;18(1):57. doi: 10.1186/s12968-016-0270-1. PMID 27624746